CLINICAL TRIAL: NCT04904068
Title: Imaging the Motor System in Parkinson's Disease
Brief Title: Functional Neuroimaging in Parkinson's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Roxana Burciu, Assistant Professor, University of Delaware
Other Study IDs: 1407867
Record Dates: First submitted 2021-02-18; First posted 2021-05-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; Healthy Aging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's disease: Individuals with a clinical diagnosis of Parkinson's disease.
- Healthy: Healthy individuals with no known neurological disorders.

SUMMARY:
The study uses magnetic resonance imaging (MRI) to better understand changes in the brain underlying motor symptoms affecting upper and lower limbs in Parkinson's disease.

DETAILED DESCRIPTION:
There is a tremendous need to improve the understanding of the pathophysiology underlying motor symptoms in Parkinson's disease in order to optimize existing treatment options/develop new therapies. This study seeks to further the understanding of impaired movement in Parkinson's disease by examining brain changes and how these relate to changes in motor behavior.

The study uses magnetic resonance imaging (MRI), a noninvasive imaging technique that does not include X-rays. MRI will assess brain activity in response to simple and coordinated movements of the upper and lower limbs that participants have to perform inside the MRI scanner. Motor and cognitive function outside the scanner using various clinical and behavioral tests will also be assessed. The study includes 1 visit to the University of Delaware.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Parkinson's disease
* No neurological disorders if interested in participating as a control participant
* Must be capable of providing informed consent
* Must be eligible to receive a brain MRI

Exclusion Criteria:

* A secondary movement disorder diagnosis in addition to Parkinson's disease
* Dementia
* Medical conditions that may make one ineligible for receiving a brain MRI
* Inability to provide informed consent
* Control/healthy group: neurological disorders
* Control/healthy group: cannot walk without an assistive device/mobility problems

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Open to local community as well as residents in DE or other nearby states willing to travel to the University of Delaware for the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Functional MRI activity during a motor task | Baseline
  Functional MRI activity during isolated/coordinated movements of the upper and lower limbs

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale | Baseline
  Only the motor section will be scored. Maximum points: 84 (the higher the score, the more severe the motor symptoms)
Kinesia One | Baseline
  Instrumented measures of motor dysfunction in Parkinson's disease. Maximum points: 72 (the higher the score, the more severe the motor symptoms)
Timed Up and Go | Baseline
  Mobility test (instrumented). Measures: duration (s), lean angle during sit/stand (degrees), turning duration (s) and turning angle (degrees)
360-Degree Turn Test | Baseline
  Instrumented test measuring dynamic balance. Measures: turning angle (degrees), turning duration (s), turning velocity (degrees/s)
Five Times Sit to Stand | Baseline
  Instrumented test measuring ability to perform transitional movements (i.e., get up from a chair). Measures: Duration (s), duration of the different phases (sitting/standing) (s), lean angle during the two phases (sitting/standing) (degrees)
The Modified Clinical Test of Sensory Interaction and Balance (mCTSIB) | Baseline
  Instrumented test assessing balance under different test conditions (eyes open/closed on firm/foam surface). Measures of postural sway: sway area (m^2/s^4), jerk (m^2/s^5), mean velocity (m/s), path length (m/s^2)
2-Minute Walking Test | Baseline.
  Instrument test assessing gait under three different conditions: 1) self-selected/normal speed, 2) self-selective/normal speed + cognitive task, 3) fast speed. Measures calculated for each condition/side of body: cadence (steps/min), double support (%GCT), gait cycle duration (s), gait speed (m/s), lateral step variability (cm), toe off angle (degrees), foot strike angle (degrees), turn velocity (degrees/s), upper limb range of motion (degrees), arm swing velocity (degrees/s).
Purdue Pegboard Test | Baseline
  Test measuring dexterity by counting the number of pegs placed on the pegboard during a given time.
Grooved Pegboard | Baseline
  Test measuring dexterity by counting how long it takes to place a given number of pegs on the pegboard.
Montreal Cognitive Assessment Test | Baseline
  Test measuring global cognitive function. Maximum points: 30 (the higher the score, the better the cognitive function)
Brief Test of Attention | Baseline
  Test measuring attention. Two sections are used that evaluate attention during reading of lists of letters and numbers. Maximum points across the two sections: 20 (the higher the score, the better the attention)
Beck Depression Inventory II | Baseline
  Questionnaire measuring depression. Maximum points: 63 (high score indicates depression)
Parkinson's Disease Questionnaire (PDQ-39) | Baseline
  Questionnaire measure health-related quality of life. Eight dimensions ranging from 0-100 (the higher the score, the worse the quality of life)
Schwab and England Activities of Daily Living Scale | Baseline
  Questionnaire on ability to complete daily task. 10% increments with 100% meaning an individual is completely independent when it comes to completing daily activities
Rapid Eye Movement Behavior Disorder Questionnaire | Baseline
  Questionnaire measuring sleep behavior. Maximum points: 13 (a high score is indicative of RBD sleep disorder)
Epworth Sleepiness Scale | Baseline
  Questionnaire measuring sleepiness. Maximum points: 24 (high score indicates sleepiness)
University of Pennsylvania Smell Identification Test | Baseline
  Test measuring sense of smell. Maximum points: 40 (the higher the score, the more normal the smell)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana G Burciu, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No